CLINICAL TRIAL: NCT05443880
Title: Multidimensional Approach (Exercise and Mindfulness) for Health Improvement in Patients With Non-specific Chronic Low Back Pain: The BackFit Project
Brief Title: Exercise and Mindfulness in Patients With Non-specific Chronic Low Back Pain: The BACKFIT Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBS Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); ISCIII (Unknown); European Social Fund (Other)
Responsible Party: Principal Investigator, Víctor Segura Jiménez, Principal Investigator, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS.Granada
Record Dates: First submitted 2022-06-02; First posted 2022-07-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: Exercise, mindfulness, sedentary behaviour, strength, pain
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain | interventions — Exercise; Mindfulness; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise (Experimental): The exercise intervention will undergo a exercise program 2 days / week (45 minutes per session) during a period of 8 weeks.
  Interventions: Behavioral: Exercise
- Exercise + mindfulness (Experimental): The exercise + mindfulness intervention will carry out a an exercise intervention together with mindfulness intervention 1 day / week (2.5 hour per session).
  Interventions: Behavioral: Exercise + mindfulness
- Control (Other): The control group will be provided with the usual care received in the Physical Medicine and Rehabilitation Service: stretching, breathing and motor control exercises 2 days / week (45 minutes per session) during a period of 8 weeks
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention will focus on working the core muscles, starting with low-intensity isometric contraction of the core muscles that stabilize the trunk; increasing intensity by performing functional tasks (phase 1: independent isometric contraction of transversus-abdominis and multifidus, phase 2: co-contraction and functional tasks of the deep trunk muscles; phase 3: functional task with load; phase 4: functional task with unstable surface)
  Arms: Exercise
Behavioral: Exercise + mindfulness — The Mindfulness Based Stress Reduction (MBSR) program will strictly follow the protocol developed by Jon Kabat Zinn. Each session will include three activities: the presentation of a topic, moments of dialogue and exploration in group (using appreciative inquiry) and a Mindfulness practice. Participants will be provided with workbooks, audios with guided meditations, and instructions for practice at home. In addition, the Exercise + mindfulness intervention will include the exercise program described in the exercise intervention.
  Arms: Exercise + mindfulness
Other: Control group — The control group will be provided with the usual care received in the Physical Medicine and Rehabilitation Service: stretching, breathing and motor control exercises 2 days / week (45 minutes per session) during a period of 8 weeks.
  Arms: Control

SUMMARY:
Chronic low back pain is among the most common health problems seen in primary care, and is responsible for disability and absenteeism in our country. In most cases, it is attributed to a non-specific cause and classified as non-specific chronic low back pain (NSCLBP). Taking into consideration that multidimensional programs usually present more effectiveness reducing pain than unimodal programs, the current research investigates the role of unexplored multidimensional program (exercise and mindfulness) in NSCLBP. The primary aim of this project is to determine the effectiveness of a supervised exercise program (intervention 1) and a supervised exercise program + mindfulness (intervention 2) on pain, disability, trunk muscle endurance/strength, quality of life and gait parameters in patients with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

* Be previously diagnosed with NSCLBP pain by a healthcare professional according to the criteria established by O'Sullivan et al.
* Intend to participate in the intervention and perform all the tests included in the study.
* Able to read and understand informed consent, as well as the objective of the study.
* Able to walk and move without outside help.
* Able to communicate without problems
* Be between 18 and 65 years old.

Exclusion Criteria:

* Having spondylolysis, spondylolisthesis, canal stenosis, degenerative disc disease, and/or disc herniation, tumor, trauma or fracture of the lumbar and lower limbs, Cauda equina syndrome, and radicular leg pain (given that spine degeneration issues are commonly present in asymptomatic individuals and increase with age, only serious lumbar structural disorders were considered).
* Having lumbar surgery as source of pain.
* Having acute or terminal illness.
* Having medical prescription that prevents the performance of the tests.
* Having injury or circumstance that makes it impossible to perform the tests correctly.
* Having other physical or mental illness that prevents participating in the intervention.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Muscular fitness at 2 months: The trunk muscle strength/endurance | Change from baseline at 2 months (Postest minus Retest)
  It will be measured with the Biering-Sørensen test and the plank test.
Change from baseline Muscular fitness at 5 months: The trunk muscle strength/endurance | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured with the Biering-Sørensen test and the plank test.
Change from baseline Muscular fitness at 2 months: lower body strength | Change from baseline at 2 months (Postest minus Retest)
  It will be measured by the 30s chair stand test. Upper body strength (maximal isometric strength) will be measured with the handgrip strength test (TKK dynamometer).
Change from baseline Muscular fitness at 5 months: lower body strength | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured by the 30s chair stand test. Upper body strength (maximal isometric strength) will be measured with the handgrip strength test (TKK dynamometer).
Change from baseline Muscular fitness at 2 months: upper body strength | Change from baseline at 2 months (Postest minus Retest)
  It will be measured with the handgrip strength test (TKK 5101 Grip-D; Takey, Tokyo, Japan dynamometer).
Change from baseline Muscular fitness at 5 months: upper body strength | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured with the handgrip strength test (TKK 5101 Grip-D; Takey, Tokyo, Japan dynamometer).

OTHER OUTCOMES:
Change from baseline Pressure pain threshold (PPT) in the lower back at 2 months | Change from baseline at 2 months (Postest minus Retest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Pressure pain threshold (PPT) in the lower back at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Disability due to pain at 2 months | Change from baseline at 2 months (Postest minus Retest)
  It will be assessed with the Oswestry low back pain scale. The total score will be calculated summing the value of the 10 items and represented as percentage (%), where 0-20% means minimum functional limitation; 20%-40% moderate functional limitation; 40%-60% intense functional limitation; 60%-80% disability and more than 80% maximum functional limitation.
Change from baseline Disability due to pain at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  It will be assessed with the Oswestry low back pain scale. The total score will be calculated summing the value of the 10 items and represented as percentage (%), where 0-20% means minimum functional limitation; 20%-40% moderate functional limitation; 40%-60% intense functional limitation; 60%-80% disability and more than 80% maximum functional limitation.
Change from baseline Pain intensity at 2 months | Change from baseline at 2 months (Postest minus Retest)
  Patients will be instructed to indicate the intensity of pain they felt on a valid and reliable 10 cm long straight line marked with a score from 0 to 10
Change from baseline Pain intensity at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  Patients will be instructed to indicate the intensity of pain they felt on a valid and reliable 10 cm long straight line marked with a score from 0 to 10
Change from baseline Sedentary time and physical activity at 2 months | Change from baseline at 2 months (Postest minus Retest)
  They will be recorded through GT3X+ Accelerometer (Actigraph, Inc., Fort Walton Beach, FL, USA).
Change from baseline Sedentary time and physical activity at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  They will be recorded through GT3X+ Accelerometer (Actigraph, Inc., Fort Walton Beach, FL, USA).
Change from baseline Gait parameters at 2 months | Change from baseline at 2 months (Postest minus Retest)
  Spatiotemporal parameters (e.g., cadence, stance and support times, step length and stride width) will be calculated using Optogait.
Change from baseline Gait parameters at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  Spatiotemporal parameters (e.g., cadence, stance and support times, step length and stride width) will be calculated using Optogait.
Change from baseline Fat percentage at 2 months | Change from baseline at 2 months (Postest minus Retest)
  will be measured by bioelectrical impedance analysis (InBody R20, Biospace)
Change from baseline Fat percentage at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  will be measured by bioelectrical impedance analysis (InBody R20, Biospace)
Change from baseline weight (kg) and height (cm) to report BMI in kg/m^2 at 2 months | Change from baseline at 2 months (Postest minus Retest)
  they will be measured by bioelectrical impedance analysis (InBody R20, Biospace) and height rod (Seca 22).
Change from baseline weight (kg) and height (cm) to report BMI in kg/m^2 at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  they will be measured by bioelectrical impedance analysis (InBody R20, Biospace) and height rod (Seca 22).
Change from baseline Health-related quality of life at 2 months | Change from baseline at 2 months (Postest minus Retest)
  will be assessed with the Short-Form Health Survey (SF-36). It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. The scores range from 0 to 100 in every dimension, where higher scores indicate better health.
Change from baseline Health-related quality of life at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  will be assessed with the Short-Form Health Survey (SF-36). It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. The scores range from 0 to 100 in every dimension, where higher scores indicate better health.
Change from baseline Central sensitization at 2 months | Change from baseline at 2 months (Postest minus Retest)
  The Central Sensitisation Inventory will be used. It is a self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitisation. It presents 25 questions and the patient scores each answer on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation
Change from baseline Central sensitization at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  The Central Sensitisation Inventory will be used. It is a self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitisation. It presents 25 questions and the patient scores each answer on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation
Change from baseline Pain Catastrophyzing at 2 months | Change from baseline at 2 months (Postest minus Retest)
  The Pain Catastrophizing Scale will be used to assess painful experiences and thoughts or feelings about pain. It contains 13 items on a 5-point scale. Higher score represents a more negative appraisal of pain.
Change from baseline Pain Catastrophyzing at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  The Pain Catastrophizing Scale will be used to assess painful experiences and thoughts or feelings about pain. It contains 13 items on a 5-point scale. Higher score represents a more negative appraisal of pain.
Change from baseline Depression severity at 2 months | Change from baseline at 2 months (Postest minus Retest)
  The Beck Depression Inventory-II will be used. It contains 21 items and the range of score is 0-63 with higher values indicating greater depression.
Change from baseline Depression severity at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  The Beck Depression Inventory-II will be used. It contains 21 items and the range of score is 0-63 with higher values indicating greater depression.
Change from baseline Anxiety state at 2 months | Change from baseline at 2 months (Postest minus Retest)
  The State Trait Anxiety Inventory-I will be used to assess anxiety state (i.e., the level of current anxiety). It is a 20-item self-administered questionnaire and the range of score is 20-80, with higher score indicating a greater anxiety state.
Change from baseline Anxiety state at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  The State Trait Anxiety Inventory-I will be used to assess anxiety state (i.e., the level of current anxiety). It is a 20-item self-administered questionnaire and the range of score is 20-80, with higher score indicating a greater anxiety state.
Change from baseline Sleep duration and quality at 2 months | Change from baseline at 2 months (Postest minus Retest)
  It will be assessed with the Pittsburgh Sleep Quality Index. It is composed of 19 questions, with four-point Likert scales (0-3), addressing seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The sleep quality global score is the sum of all components. Higher scores indicate worse sleep quality.
Change from baseline Sleep duration and quality at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  It will be assessed with the Pittsburgh Sleep Quality Index. It is composed of 19 questions, with four-point Likert scales (0-3), addressing seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The sleep quality global score is the sum of all components. Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- IBS.Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No